CLINICAL TRIAL: NCT06486116
Title: Effectiveness of Task Specific Home Exercise Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York Presbyterian Brooklyn Methodist Hospital (Other)
Responsible Party: Principal Investigator, Karen Blitz-Shabbir, Neurologist, New York Presbyterian Brooklyn Methodist Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2160034
Record Dates: First submitted 2024-06-21; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized Task Specific Physical Therapy Home Exercise Program (Experimental): Physical Therapy Home Exercise program based on specific outcome measure findings.
  Interventions: Behavioral: Task Specific Physical Therapy Home Program
- Generic physical therapy home exercise program (Active Comparator): Generalized fitness-based exercise program
  Interventions: Behavioral: Task Specific Physical Therapy Home Program

INTERVENTIONS:
Behavioral: Task Specific Physical Therapy Home Program — Home exercise program based on specific findings from physical therapy evaluations.

SUMMARY:
The purpose of this study is to compare the effectiveness of 2 different types of Home Exercise Programs (HEP) on mobility in persons with Multiple Sclerosis (MS). Specifically, we will be comparing the Standard of Care (SOC) a program based on aerobic conditioning and calisthenics to a Task Specific Program (TSP).

Primary Question: Will persons with who receive a Task Specific HEP have greater improvement in mobility than those who receive the SOC? Secondary question: Will a task specific HEP be as well tolerated as the SOC HEP by persons with MS

DETAILED DESCRIPTION:
Persons with MS have been shown to benefit from exercise to address the symptoms of their disease. Exercise programs are customarily given by Physical Therapists (PT) in either an inpatient or outpatient setting. Outpatient PT is typically augmented with a Home exercise Program (HEP) which is meant to enhance the work that is done directly with the PT. Since the amount of exercise done at home is often greater than what is done with the PT, the HEP is of great importance.

However, the types of exercise that are the most useful for useful for persons with MS has not been established. Previous research has shown that due to the unique ways in which MS can affect the nervous system, exercise programs that may be appropriate for persons without MS may not be ideal for those that have the disease

ELIGIBILITY:
Inclusion Criteria:

Definitive diagnosis of Multiple sclerosis

* Ability to walk for at least 30 seconds unassisted with or without assistive device
* Ability to read, comprehend and sign an informed consent
* Is able to attend a 2 outpatient evaluation sessions 6 weeks apart
* Between the ages of 18 and 75

Exclusion Criteria:

* Evidence of recent MS exacerbation

  * Any orthopedic, cardiopulmonary, or non- MS neurologic condition that prohibits participation in a Physical therapy program
  * Be currently receiving outpatient physical therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
6 Minute Walk Test | Measured before and after each 4 weeks
  Participant walks at best comfortable pace for 6 consecutive minutes; total distance walked and distance per minute is measured.
The Functional Gait Assessment | Measured before and after each 4 weeks
  A measure of walking balance assessed by participant's performance on specific task.
The Mini Balance Evaluation Systems Test (MBEST) | Measured before and after each 4 weeks
  Assessment of participant balance during reactive anticipatory, dynamic and sensory aspects of balance tasks.

CONTACTS AND LOCATIONS:
Locations (1):
- New York Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available. The specific individual participant data sets are to be shared are, collected IPD, all IPD that underlie results in a publication.
Supporting Information: Study Protocol
Time Frame: Data will be shared following publication of our findings in an article in the appropriate peered review journal.
Access Criteria: Requests for data will be considered on an individual basis by the Principal Investigator.

REFERENCES:
- [Background] Ghahfarrokhi MM, Banitalebi E, Negaresh R, Motl RW. Home-Based Exercise Training in Multiple Sclerosis: A Systematic Review with Implications for Future Research. Mult Scler Relat Disord. 2021 Oct;55:103177. doi: 10.1016/j.msard.2021.103177. Epub 2021 Jul 27. PMID 34343867
- [Background] Dalgas U, Ingemann-Hansen T, Stenager E. Physical Exercise and MS Recommendations. Int MS J. 2009 Apr;16(1):5-11. PMID 19413920
- [Background] Ozkul C, Guclu-Gunduz A, Eldemir K, Apaydin Y, Gulsen C, Yazici G, Soke F, Irkec C. Effect of task-oriented circuit training on motor and cognitive performance in patients with multiple sclerosis: A single-blinded randomized controlled trial. NeuroRehabilitation. 2020;46(3):343-353. doi: 10.3233/NRE-203029. PMID 32310197
- [Background] McGuigan C, Hutchinson M. The multiple sclerosis impact scale (MSIS-29) is a reliable and sensitive measure. J Neurol Neurosurg Psychiatry. 2004 Feb;75(2):266-9. PMID 14742602
- [Background] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Background] Goldman MD, Ward MD, Motl RW, Jones DE, Pula JH, Cadavid D. Identification and validation of clinically meaningful benchmarks in the 12-item Multiple Sclerosis Walking Scale. Mult Scler. 2017 Sep;23(10):1405-1414. doi: 10.1177/1352458516680749. Epub 2016 Dec 7. PMID 27903937
- [Background] Savci S, Inal-Ince D, Arikan H, Guclu-Gunduz A, Cetisli-Korkmaz N, Armutlu K, Karabudak R. Six-minute walk distance as a measure of functional exercise capacity in multiple sclerosis. Disabil Rehabil. 2005 Nov 30;27(22):1365-71. doi: 10.1080/09638280500164479. PMID 16372431
- [Background] Forsberg A, Andreasson M, Nilsagard Y. The Functional Gait Assessment in People with Multiple Sclerosis: Validity and Sensitivity to Change. Int J MS Care. 2017 Mar-Apr;19(2):66-72. doi: 10.7224/1537-2073.2015-061. PMID 32607064
- [Background] Potter K, Bowling R, Kavanagh L, Stone A, Witt B, Wooldridge A. Reliability, Validity, and Responsiveness of the Mini-Balance Evaluation Systems Test in Ambulatory Individuals with Multiple Sclerosis. Physiother Can. 2019 Fall;71(4):327-334. doi: 10.3138/ptc-2018-0071. PMID 31762543